CLINICAL TRIAL: NCT01507597
Title: The Effect of GLP-1 on the Inhibition of Glucagon Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, Principal Investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GlukaStase; H-3-2011-088 (Other: The Danish National Committee for Research Ethics)
Record Dates: First submitted 2011-12-13; First posted 2012-01-11 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes; Type 1 Diabetes
Keywords: Glucagon-like peptide-1; Glucagon; Normal physiology; T2DM; T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — glucagon-like peptide 1 (7-36)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Subjects (Other)
  Interventions: Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)); Drug: NaCl
- T2DM (Other)
  Interventions: Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)); Drug: NaCl
- T1DM (Other)
  Interventions: Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)); Drug: NaCl

INTERVENTIONS:
Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)) — Continuous iv. infusion of the native gut hormone GLP-1 (0.2 pmol/kg/min) for 210 minutes.
  Combined with a step wise glucose clamp using 20% w/w glucose iv. infusion reaching plasma glucose value of 15 mM starting at fasting plasma glucose (30 min per step)
Drug: NaCl — Continuous iv. saline infusion (NaCl Isotonic) for 210 minutes. Combined with a step wise glucose clamp using 20% w/w glucose iv. infusion reaching plasma glucose value of 15 mM starting at fasting plasma glucose (30 min per step)
Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)) — Continuous iv. infusion of the native gut hormone GLP-1 (0.4 pmol/kg/min) for 210 minutes.
  Combined with a step wise glucose clamp using 20% w/w glucose iv. infusion reaching plasma glucose value of 15 mM starting at fasting plasma glucose (30 min per step)
Drug: Native human Glucagon-like Peptide-1 ( GLP-1(7-36)) — Continuous iv. infusion of the native gut hormone GLP-1 (0.8 pmol/kg/min) for 210 minutes.
  Combined with a step wise glucose clamp using 20% w/w glucose iv. infusion reaching plasma glucose value of 15 mM starting at fasting plasma glucose (30 min per step)

SUMMARY:
Diabetes(both types) are recognized by high levels of glucagon in the circulation.

Glucagon is known to increase blood glucose, and might therefore contribute to the respective diseases. Under some circumstances the gut hormone GLP-1 inhibits the glucagon secretion.

The investigators aim to identify the impact of GLP-1 on the glucagon secretion, at increasing blood glucose levels in healthy subjects, in patients with type 2 diabetes, and in patients with type 1 diabetes.

The investigators think that the effect of GLP-1 on the glucagon secretion might be dependent of blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

Patients with T2DM

* Above the age of 35 years, treatment with diet or oral anti-diabetic medication. Diagnosed with T2DM in at leat three months in advance(WHO criterion)
* Normal hemoglobin
* Informed content Patients with T1DM
* T1DM (WHO criterion)
* Plasma-C-peptid negative due to arginin-test
* Normal hemoglobin
* age> 18 years
* Informed content Healthy subjects
* Normal fasting plasma glucose and normal glucose tolerance (WHO criterion)
* Normal hemoglobin
* Age >18 years
* Informed content

Exclusion Criteria:

Patients with T2DM

* Treatment with glitazones and/or gliptins
* Inflammatory bowels disease
* previous bowel resection with or without stomy
* Nephropathy (serum creatinin >150 µM and/or albuminuria)
* Liver disease (serum alanine-aminotransferase (ALAT) and/or serum aspartate-aminotransferase (ASAT) >2×normal values)
* Medical treatment impossible to break for 12h.
* Age >80 years Patients with T1DM
* Overweight (BMI >30 kg/m2)
* Inflammatory bowels disease
* previous bowel resection with or without stomy
* Nephropathy (serum creatinin >150 µM and/or albuminuria)
* Liver disease (serum alanine-aminotransferase (ALAT) and/or serum aspartate-aminotransferase (ASAT) >2×normal values)
* Medical treatment impossible to break for 12h (except treatment with insulin).
* Age >80 years

Healthy subjects

* Diabetes
* Prediabetes (impaired glucose tolerance and/or impaired fasting plasma glucose)
* First order relatives with diabetes
* Overweight (BMI >30 kg/m2)
* Inflammatory bowels disease
* previous bowel resection with or without stomy
* Nephropathy (serum creatinin >150 µM and/or albuminuria)
* Liver disease (serum alanine-aminotransferase (ALAT) and/or serum aspartate-aminotransferase (ASAT) >2×normal values)
* Medical treatment impossible to break for 12h.
* Age >80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Plasma Glucagon response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  The collection of blood samples will be done during the 210 min GLP-1 infusion / glucose clamp-session
Plasma GLP-1 response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  The collection of blood samples will be done during the 210 min GLP-1 infusion / glucose clamp-session
Plasma Glucose response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  The collection of blood samples will be done during the 210 min GLP-1 infusion / glucose clamp-session

SECONDARY OUTCOMES:
Resting Metabolic Rate response to the GLP-1 infusion / glucose clamp | at 0, 120, and 180 min
  Assessed by indirect calorimetry during the GLP-1 infusion / glucose clamp-session
Hunger scores response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  Assessed by VAS during the 210 min GLP-1 infusion / glucose clamp-session
plasma Insulin response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  The collection of blood samples will be done during the 210 min GLP-1 infusion / glucose clamp-session
plasma GIP response to the GLP-1 infusion / glucose clamp | At 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210 min
  The collection of blood samples will be done during the 210 min GLP-1 infusion / glucose clamp-session
Food Intake | at 210 min
  Assessed by ad'libitum meal after the 210 min GLP-1 infusion / glucose clamp.

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Bagger JI, Grondahl MFG, Lund A, Holst JJ, Vilsboll T, Knop FK. Glucagonostatic Potency of GLP-1 in Patients With Type 2 Diabetes, Patients With Type 1 Diabetes, and Healthy Control Subjects. Diabetes. 2021 Jun;70(6):1347-1356. doi: 10.2337/db20-0998. Epub 2021 Mar 15. PMID 33722838